CLINICAL TRIAL: NCT05670080
Title: Does Motor Imagination Have a Therapeutic Role in Arthroscopic Rotator Cuff Repair? Randomized Controlled, Single-Blind Trial
Brief Title: Does MI Have a Therapeutic Role in Arthroscopic Rotator Cuff Repair?
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the continuation of my PhD thesis process, patient admission will begin after the completion of my PhD graduation.
Sponsor: Alanya Alaaddin Keykubat University (Other)
Collaborators: Pamukkale University (Other); Alanya Allaaddin Keykubat University Hospital (Unknown); Alanya Hamdullah Emin Pasha University (Unknown)
Responsible Party: Principal Investigator, Ozum Cetinkaya, Principal Investigator, Alanya Alaaddin Keykubat University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MIafterARCR
Record Dates: First submitted 2022-12-08; First posted 2023-01-04 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Rotator Cuff Tears; Motor Imagery; Muscle Activity; Atrophy, Muscular; Patient Satisfaction; Kinesiophobia; Shoulder Pain
Keywords: Motor Imagery; Muscle Activity; Muscular Atrophy; Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries; Muscular Atrophy; Patient Satisfaction; Kinesiophobia; Shoulder Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: The study will be divided into two parallel groups: the MI group and the Control group. Both groups will participate in a routine physical therapy program after 4 weeks of immobilization, with the MI group receiving additional motor imagery training during the preoperative period. MI training will be provided to Group 1 participants who are planning for rotator cuff repair in the pre-surgical period by the corresponding researcher. The physical therapy program will be applied by a physiotherapist with a master's degree and 8 years of professional experience in the field of orthopedic rehabilitation, who is different from the corresponding researcher of the study.
Who Masked: Participant, Care Provider
Masking Description: A physiotherapist with a master's degree who is unaware of the study's content will apply the physical therapy program and assessments.
  Participants will take physical therapy program and MI training without being told which group they were in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Motor Imagery (MI) Group (Experimental): MI training will be prepared using the Microsoft PowerPoint program which includes written, visual and audio materials, as well as features that can be sent to participants ' phones/tablets/computers. The MI training will allow the participant to perform visual and kinesthetic imagery with visual and audible notifications and will include 6 exercises for the muscles around the shoulder, 3 exercises for strengthening, and dynamic stabilization for the muscles around the scapula. In each presentation, verbal cues will be given to explain how to imagine the movement while a visual of the motor movement is displayed on the screen. During MI exercises, participants will be called once a week and their MI practices will be followed up.
  After the first four weeks of MI training, the MI group will also participate in a four-week physical therapy program.
  Interventions: Behavioral: Motor Imagery; Behavioral: Physical Therapy
- Physical Therapy (PT) Group (Experimental): Following the preoperative evaluations, both groups will be shown remedial exercises (pumping exercises that activate the circulation), flexion, and extension wrist exercises, which they should do for four weeks.
  After a 4-week immobilization period, participants in the PT Group will begin a physical therapy program that includes routine electrotherapy (TENS), cold pack therapy, joint range of motion exercises, and strengthening exercises for the muscles around the shoulder.
  Interventions: Behavioral: Physical Therapy

INTERVENTIONS:
Behavioral: Motor Imagery — Motor imagery is the imagining of action without its physical execution and motor imagery elicits activity in brain regions that are normally activated during actual task performance. The brain perceives real experiences and the visualization process as similar. For this reason, imagery is considered a mental exercise
  Arms: The Motor Imagery (MI) Group
Behavioral: Physical Therapy — Electrotherapy (TENS), cold pack therapy, joint range of motion exercises, and strengthening exercises for the muscles around the shoulder.

SUMMARY:
Objective: The aim of this study is to investigate the effect of motor imagery on muscle activity, pain, and function in arthroscopic rotator cuff repair.

Methods: As a result of the power analysis (G-Power), 36 participants are planned to be included in this study Block randomization will be used to divide participants into 2 groups, each with at least 18 participants: Group 1 (MI group) and Group 2 (Control group) (Randomizer.org). Both groups will receive a 4-week physical therapy program. MI (Motor Imagination) group will receive a motor imagination program in addition to the physical therapy program. Data will collect using the visual analog scale (VAS), goniometric measurement, circumference measurement, Disabilities of the Arm, Shoulder, and Hand Questionnaire (DASH), Kinesthetic and Visual Imagery Questionnaire- KVIQ-20, Tampa Kinesiophobia Scale, 3-question satisfaction questionnaire, superficial Electromyography (EMG) (BTS Bioengineering Free EMG 100 RT).

Practice Implications: The current study will contribute to understanding how motor imagination affects muscle activity and muscle atrophy.

DETAILED DESCRIPTION:
After shoulder trauma, the rotator cuff may sustain tears of varying degrees. Degenerative rotator cuff tears are an important cause of shoulder pain and dysfunction. Rotator cuff injuries can be treated conservatively, medically, and surgically. Surgical treatment can be performed as arthroscopic-assisted mini-open or full arthroscopic techniques. After rotator cuff repair, long-term immobilization can lead to complications of scar formation and related shoulder stiffness, pain, muscle/tendon atrophy, and delayed return to functional and occupational activities. Motor imagery (MI) can be used in cases that cause immobilization such as pain, fatigue, and loss of strength during and after injury, or in cases of limited access to healthcare facilities.

Motor imagery is the imagining of action without its physical execution and motor imagery elicits activity in brain regions that are normally activated during actual task performance. The brain perceives real experiences and the visualization process as similar. For this reason, imagery is considered a mental exercise. The functional equivalence hypothesis shows that there is a great deal of overlap between the neural substrates of physical and imagined movement execution.

In a study examining brain signals during magnetoencephalographic (MEG) evaluation and motor movements, it was stated that the primary motor (less than motor activity) and posterior parietal cortex were activated during MI.

Today, the majority of mental exercise studies are carried out in the field of neurological rehabilitation. There are many studies on stroke, multiple sclerosis, Parkinson's, spinal cord injury, and phantom pain. MI is an effective method for motor learning that is also used in orthopedics and sports. The MI application may be an appropriate tool for professional athletes to maintain and improve their physical performance capacity. In a systematic review of the effect of MI on pain and motor function after spinal cord injury, the majority of the findings confirmed the benefits of MI interventions on the motor function when used concurrently with physical exercises. According to the findings of the systematic review published by Colmenero et al., MI has positive effects on phantom pain. Studies in patients with chronic shoulder pain syndrome and subacromial impingement syndrome have reported positive effects of MI on pain and shoulder function and active range of motion. Significantly positive results were observed in pain and disability scores after the 4th week with MI application in rotator cuff patients. Significantly positive results were observed in pain and disability scores after the 4th week of MI application in rotator cuff patients. In conclusion, extensive experimental research indicates that MI is a valuable and cost-effective technique for improving engine performance and recovery. There has been no research into the effectiveness of MI after rotator cuff repair.

The aim of this study is to investigate the effect of motor imagery on muscle activity, pain, and function in arthroscopic rotator cuff repair.

Methods:

Participants:

Volunteer participants who applied to the Orthopedics and Traumatology unit at Alanya Alaaddin Keykubat University Hospital, underwent arthroscopic rotator cuff repair by the same surgeon, and met the inclusion and exclusion criteria will take part in the study. Each participant enrolled in the study will be given detailed information about the study, and their written and verbal consent will be obtained.

According to the power analysis made with the G-power program, it was found that 80% power can be obtained with 95% confidence when at least 30 people are included in the study. While calculating the sample size, the results of the superficial EMG (-superior trapezius muscle peak dynamic value [experimental group: 35.99 (standard deviation: 14.39), control group 19.57 (standard deviation: 15.97)] were taken as a basis, and the effect size was calculated as = 1.08. The risk of case loss was taken into account by taking a reserve rate of 20%, and it was planned to include 36 participants. The cases will be divided into 2 groups by block randomization using the internet program, consisting of at least 18 individuals: Group 1 [MI group] and Group 2 [Control group] (Randomizer.org).

Study Protocol:

The study will be divided into two parallel groups: the MI group and the Control group. Both groups will participate in a routine physical therapy program after 4 weeks of immobilization, with the MI group receiving additional motor imagery training during the preoperative period.

A physiotherapist with a master's degree who will apply for the treatment program and is unaware of the study's content will administer the assessments in the pre-operative period and post-operative 8th week. Data will collect using the descriptive Information form (prepared by the principal investigator), visual analog scale (VAS), goniometric measurement, circumference measurement, Disabilities of the Arm, Shoulder, and Hand Questionnaire (DASH), Kinesthetic and Visual Imagery Questionnaire- KVIQ-20, Tampa Kinesiophobia Scale, 3-question satisfaction questionnaire, superficial Electromyography (EMG) (BTS Bioengineering Free EMG 100 RT).

Training and Exercise Applications:

MI training will be provided to Group 1 participants who are planning for rotator cuff repair in the pre-surgical period. The training will be prepared using the Microsoft PowerPoint program which includes written, visual and audio materials, as well as features that can be sent to participants ' phones/tablets/computers.

MI training will allow the participant to perform visual and kinesthetic imagery with visual and audible notifications and will include 6 exercises for the muscles around the shoulder, 3 exercises for strengthening, and dynamic stabilization for the muscles around the scapula. In each presentation, verbal cues will be given to explain how to imagine the movement while a visual of the motor movement is displayed on the screen. Participants will be given 10 seconds of time, beginning and ending with an audible beep, and each exercise will be repeated 10 times before transitioning to the next exercise. Participants will be told in detail that they should begin MI exercises on the third day after surgery and continue them for four weeks. During MI exercises, participants will be called once a week and their MI practices will be followed up, as well as support for the questions and problems they experience. Group 1 will then participate in a 4-week physical therapy program, which will include electrotherapy, cold application, joint range of motion exercises, and strengthening exercises for the muscles around the shoulder.

Following the preoperative evaluations, both groups will be shown remedial exercises (pumping exercises that activate the circulation), flexion, and extension wrist exercises, which they should do for four weeks. After a 4-week immobilization period, participants in Group 2 will begin a physical therapy program that includes routine electrotherapy (TENS), cold pack therapy, joint range of motion exercises, and strengthening exercises for the muscles around the shoulder. The MI training will be applied by the principal investigator. The physical therapy program will be applied by a physiotherapist with a master's degree and 8 years of professional experience in the field of orthopedic rehabilitation, who is different from the principal investigator of the study.

Statistical Analysis:

In the statistical analysis of data will obtain in this study, a Windows-based SPSS (IBM SPSS Statistics, Version 24.0, Armonk, NY, USA) package program will use. Continuous variables will express as a mean ± standard deviation or as a median (minimum-maximum values), and categorical variables as a number and percent. Analytical (Kolmogorov-Smirnov/Shapiro-Wilks test) and visual (Histogram and probability graphs) methods will use to test the conformity of data for normal distribution. When the parametric test assumptions were provided, Independent Sample T-Test will use to compare independent group differences; when the parametric test assumptions were not provided, the Mann Whitney-U test will use to compare independent group differences. In the dependent group analyses; when the parametric test assumptions were provided, Paired Sample T-Test will use; when the parametric test assumptions were not provided, Wilcoxon Test will use. Chi-Square Analysis and Fisher Exact Test will use compare differences between categorical variables.

ELIGIBILITY:
Inclusion Criteria:

* Ability to speak and understand Turkish - Previous arthroscopic rotator cuff repair
* Achieving a minimum of 40 points on the Kinesthetic and Visual Imagery Questionnaire -20 (KGIA-20)
* Access to adequate technological devices for communication and follow-up

Exclusion Criteria:

* Who with neurological diseases that may cause functional impairment.
* Patients who have another shoulder problem and/or have had previous shoulder surgery on the same upper extremity.
* Who wanted to leave the study at their own request
* Who could not continue to work due to any additional discomfort developed

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-09-15 (Estimated); Primary Completion 2027-07-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Change of Muscle activity | 1 week before surgery and week 8 after surgery
  Change of Muscle activity will be evaluated with superficial Electromyography (EMG) (BTS Bioengineering Free EMG 100 RT).
Change of shoulder functional level | 1 week before surgery and week 8 after surgery
  Disabilities of the Arm, Shoulder, and Hand Questionnaire (DASH) will be used to determine the upper extremity functional level.The total of all item scores was then used to calculate the interrogation score, which ranged from 0 (no disability) to 100. (most severe disability). The first 20 questions concern physical competence, while the last ten concern pain and functional and environmental limitations.
Change of Kinesthetic and visual imagery levels | 1 week before surgery and week 8 after surgery
  The Kinesthetic and Visual Imagery Questionnaire- KVIQ-20 will be used to assess the kinesthetic and visual imagery levels of healthy and physically disabled individuals.The questionnaire contains a total of 20 titles, 10 of which are visual and 10 of which are kinesthetic. The intensity level of imagery is recorded on a 5-point Likert scale with the questionnaire (5 = appearance of a live image; 1 = no image or sensation).
Change of Kinesiophobia | 1 week before surgery and week 8 after surgery
  Kinesiophobia was evaluated with Tampa Scale of Kinesiophobia (TSK).TSK is a 17-question checklist. The scale employs a 4-point Likert scoring system (1= strongly disagree, 4= completely agree).
Change of Patient Satisfaction | 1 week before surgery and week 8 after surgery
  A Numerical Evaluation Scale will be used to evaluate a 2-question satisfaction questionnaire. This scale is made up of a horizontal straight line 10 cm long. The line has a value of 0 at the start and a value of 10 at the end, from left to right. On a scale of 0 to 10, patients will be asked to rate their level of satisfaction.

SECONDARY OUTCOMES:
Descriptive Information | 1 week before surgery
  Age, gender, dominant hand, previous diseases, occupation and contact information of the patients were recorded in the descriptive information form.
Change in Pain-Visual analog scale | 1 week before surgery, week 4 and week 8 after surgery
  Pain of patients during sleep, rest and activity will evaluate using a visual analog scale (VAS).This scale is made up of a 10 cm horizontal straight line. When viewed from left to right, a 0 at the start of the line indicates no pain, and a 10 at the end indicates severe pain.
Change of Range of Motion | 1 week before surgery, week 4 and week 8 after surgery
  The limitation of shoulder joint flexion, extension, abduction, adduction, internal and external rotation movements will be measured using a universal goniometer and recorded in degrees(˚).
Change in muscle atrophy | 1 week before surgery and week 8 after surgery
  For changes in muscle atrophy, circumference measurements (one of Anthropometric measurements) will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Özüm ÇETİNKAYA EREN, PT, MSc, Principal Investigator — Alanya Alaaddin Keykubat University; Ummuhan BAŞ ASLAN, Prof.Dr.PT., Study Director — Pamukkale University; Kazım Emre EREN, PT, MSc, Study Chair — Alanya Alaaddin Keykubat University Hospital; Anıl GÜLCÜ, Asst.Prof.Dr, Study Chair — Alanya Alaaddin Keykubat University; Erdem DEMİR, Asst.Prof.Dr, Study Chair — Alanya Hamdullah Emin Paşa University
Locations (1):
- Alanya Alaaddin Keykubat University, Alanya, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Araya-Quintanilla F, Gutierrez-Espinoza H, Jesus Munoz-Yanez M, Rubio-Oyarzun D, Cavero-Redondo I, Martinez-Vizcaino V, Alvarez-Bueno C. The Short-term Effect of Graded Motor Imagery on the Affective Components of Pain in Subjects with Chronic Shoulder Pain Syndrome: Open-Label Single-Arm Prospective Study. Pain Med. 2020 Oct 1;21(10):2496-2501. doi: 10.1093/pm/pnz364. PMID 32003812
- [Background] Guillot A, Collet C, Nguyen VA, Malouin F, Richards C, Doyon J. Brain activity during visual versus kinesthetic imagery: an fMRI study. Hum Brain Mapp. 2009 Jul;30(7):2157-72. doi: 10.1002/hbm.20658. PMID 18819106
- [Background] Boden-Albala B, Roberts ET, Bazil C, Moon Y, Elkind MS, Rundek T, Paik MC, Sacco RL. Daytime sleepiness and risk of stroke and vascular disease: findings from the Northern Manhattan Study (NOMAS). Circ Cardiovasc Qual Outcomes. 2012 Jul 1;5(4):500-7. doi: 10.1161/CIRCOUTCOMES.111.963801. Epub 2012 Jul 10. PMID 22787063
- [Background] Chholak P, Niso G, Maksimenko VA, Kurkin SA, Frolov NS, Pitsik EN, Hramov AE, Pisarchik AN. Visual and kinesthetic modes affect motor imagery classification in untrained subjects. Sci Rep. 2019 Jul 8;9(1):9838. doi: 10.1038/s41598-019-46310-9. PMID 31285468
- [Background] Hayes K, Walton JR, Szomor ZR, Murrell GA. Reliability of five methods for assessing shoulder range of motion. Aust J Physiother. 2001;47(4):289-94. doi: 10.1016/s0004-9514(14)60274-9. PMID 11722295
- [Background] Matlak S, Andrews A, Looney A, Tepper KB. Postoperative Rehabilitation of Rotator Cuff Repair: A Systematic Review. Sports Med Arthrosc Rev. 2021 Jun 1;29(2):119-129. doi: 10.1097/JSA.0000000000000310. PMID 33972488
- [Background] Opsommer E, Chevalley O, Korogod N. Motor imagery for pain and motor function after spinal cord injury: a systematic review. Spinal Cord. 2020 Mar;58(3):262-274. doi: 10.1038/s41393-019-0390-1. Epub 2019 Dec 13. PMID 31836873
- [Background] Herrador Colmenero L, Perez Marmol JM, Marti-Garcia C, Querol Zaldivar MLA, Tapia Haro RM, Castro Sanchez AM, Aguilar-Ferrandiz ME. Effectiveness of mirror therapy, motor imagery, and virtual feedback on phantom limb pain following amputation: A systematic review. Prosthet Orthot Int. 2018 Jun;42(3):288-298. doi: 10.1177/0309364617740230. Epub 2017 Nov 20. PMID 29153043